CLINICAL TRIAL: NCT01483365
Title: The Use of Luteal Support After NC-FET
Brief Title: The Need for Luteal Support in NC-FET
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0087-11-WOMC-
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Abnormal Menstrual Cycle
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vaginal tablet Endometrin twice a day — Endometrin 100 mg twice a day
  Other Names: Endometrin 100 mg twice a day

SUMMARY:
The investigators are going to examine prospectively the need of luteal support after NC-FET.

DETAILED DESCRIPTION:
The investigators are going to examine retroprospectively the need of luteal support after NC-FET in IVF cycle. One arm will receive luteal support after NC FET with vaginal tablet of Endometrin 100 mg twice a day after ET. The second arm will not. We are going to evaluate the pregnancy and implantation rate.

ELIGIBILITY:
Inclusion Criteria:

* Women under 39 years old, regular menstruation going through IVF NC-FET

Exclusion Criteria:

* NO

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 4 weeks
  We would like to investigate whether there is need for luteal support in NC-FET cycle.

CONTACTS AND LOCATIONS:
Overall Officials: David Levran, M.D, Principal Investigator — IVF Unit, Department of Obstetrics and Gynecology,Wolfson Medical Center . Holon, Israel
Locations (1):
- Wolfson medical center, Holon, Israel

REFERENCES:
- [Derived] Horowitz E, Mizrachi Y, Finkelstein M, Farhi J, Shalev A, Gold E, Raziel A, Weissman A. A randomized controlled trial of vaginal progesterone for luteal phase support in modified natural cycle - frozen embryo transfer. Gynecol Endocrinol. 2021 Sep;37(9):792-797. doi: 10.1080/09513590.2020.1854717. Epub 2020 Dec 14. PMID 33307906